CLINICAL TRIAL: NCT01822912
Title: Evaluation of a Skilled Nursing Facility Heart Failure Disease Management Program Versus Usual Care
Brief Title: Heart Failure Management Program Versus Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-0006; R01HL113387 (NIH)
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Failure; Congestive Heart Failure
Keywords: Skilled Nursing Facility; Heart Failure; Transitional Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heart Failure Disease Management Program (Active Comparator): Patients will receive personalized care to include medication titration, daily weights, symptom and activity assessment, documentation of ejection fraction, patient and caregiver education,dietary surveillance, discharge instructions and follow up visit within 7 days of SNF discharge
  Interventions: Other: Heart Failure Disease Management Program
- Heart Failure Usual Care (Placebo Comparator): SNF patients with HF will receive usual care
  Interventions: Other: Heart Failure Usual Care

INTERVENTIONS:
Other: Heart Failure Disease Management Program — Subjects will be assessed 3 times a week while in SNF.
  Arms: Heart Failure Disease Management Program
Other: Heart Failure Usual Care — Subjects will receive standard of care.
  Arms: Heart Failure Usual Care

SUMMARY:
Heart Failure (HF) patients discharged to Skilled Nursing Facilities have higher rehospitalization rates and mortality than patients discharged to home.

HF disease management programs have been shown to reduce rehospitalizations in community settings, no national guidelines have been set forth for Skilled Nursing Facilities (SNF).

This study will investigate the the effect of a heart failure-disease management program on the outcome of all-cause hospital readmissions, emergency room admissions and mortality for 30 days post-SNF admission using 7 component heart failure disease management program.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure is listed as the hospital discharge primary diagnosis
* Heart Failure is listed as the hospital discharge secondary diagnosis

Exclusion Criteria:

* Any life threatening condition which predicts mortality in 6 months or less

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2013-01; Primary Completion 2018-05 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in 60 day post SNF admission outcomes | Up to 60 days post SNF admission
  To determine the difference in the composite endpoint of 60-day all-cause hospitalization, all-cause emergency department visits and all-cause mortality between HF patients in Skilled Nursing Facilities cared for by a heart failure-disease management program vs usual care.

SECONDARY OUTCOMES:
Difference in health status and self-care 60 days post SNF admission | 60 days post SNF admission
  To compare the difference in health status and self-care for patients with HF cared for by a SNF heart failure-disease management program vs usual care 60 days post SNF admission. Health Status will be measured by the KCCQ (Kansas City Cardiomyopathy Questionnaire) which is a 23 item questionnaire specific for patients with HF. It includes aspects of physical function, symptoms (frequency, severity and stability), social function, self-efficacy, knowledge, and quality of life. HF Self Management will be measured using the SCHFI (Self-Care HF Index) which consists of 15 item scale with 3 domains of self care including self care maintenance (behaviors to maintain clinical stability), self-care management (decision making process with regard to symptom changes), and confidence to manage symptoms.
Change in Patients living at home 60 days post-SNF admission with Heart Failure (HF) | 60 days post SNF admission
  To determine if a SNF HF disease management program vs. usual care results in a greater proportion of HF patients who were previously living at home return home vs. admission to long term care post SNF discharge.
Difference in Cost-effectiveness | Up to 60 days post SNF admission
  To assess the cost-effectiveness of heart failure disease management program vs usual care for SNF patients with HF

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Boxer, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lum H, Obafemi O, Dukes J, Nowels M, Samon K, Boxer RS. Use of Medical Orders for Scope of Treatment for Heart Failure Patients During Postacute Care in Skilled Nursing Facilities. J Am Med Dir Assoc. 2017 Oct 1;18(10):885-890. doi: 10.1016/j.jamda.2017.05.021. Epub 2017 Jul 6. PMID 28688730